CLINICAL TRIAL: NCT02744495
Title: Prophylaxis of Postoperative Nausea and Vomiting After Cardiac Surgery (PONVACS)
Brief Title: Prophylaxis of Postoperative Nausea and Vomiting After Cardiac Surgery
Acronym: PONVACS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hôpital Privé de Parly II - Le Chesnay (Other)
Responsible Party: Principal Investigator, Sébastien CHAMPION, Dr, Hôpital Privé de Parly II - Le Chesnay
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-A01440-49
Record Dates: First submitted 2016-04-08; First posted 2016-04-20 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Postoperative Vomiting; Postoperative Nausea; Postoperative Emesis
Keywords: cardiac surgery; corticoids; droperidol; antiemetics; Postoperative Vomiting; Postoperative Nausea; Postoperative Emesis; prophylaxis
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Betamethasone; Droperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- postoperative nausea and vomiting risk factors (Experimental): Preoperative collection of postoperative nausea and vomiting risk factors available for practicians.
  Interventions: Drug: Betamethasone; Drug: Droperidol
- control (No Intervention): No prophylaxis whatever risk score is. Postoperative nausea and vomiting risk factors not available for practicians.

INTERVENTIONS:
Drug: Betamethasone — Prophylaxis if risk score is over 2. Prophylaxis of postoperative nausea and vomiting by betamethasone / Celestene (4mg) and/or droperidol / Droleptan (0.625mg) immediately after cardiac surgery, depending on risk factors in the intervention arm.
  Other Names: Celestene
  Arms: postoperative nausea and vomiting risk factors
Drug: Droperidol — Prophylaxis if risk score is over 2. Prophylaxis of postoperative nausea and vomiting by betamethasone / Celestene (4mg) and/or droperidol / Droleptan (0.625mg) immediately after cardiac surgery, depending on risk factors in the intervention arm.
  Other Names: Droleptan
  Arms: postoperative nausea and vomiting risk factors

SUMMARY:
To investigate the role of postoperative nausea and vomiting risk factors assessment after cardiac surgery. We designed a randomized controlled study comparing standard care (no risk factor assessment and no intervention) with prophylaxis of postoperative nausea and vomiting after cardiac surgery in high risk patients. Prophylaxis of postoperative nausea and vomiting by betamethasone (4mg) and/or droperidol (0.625mg) immediately after cardiac surgery, depending on risk factors (if risk score is over 2) in the intervention arm.

DETAILED DESCRIPTION:
Patients planned to undergo cardiac surgery were screened for inclusion. Inclusion criteria are as follow: Non emergent cardiac surgery; Age > 18 years; Affiliation to French Social Security; Approval of participation to the study; at the exclusion of: Pregnancy ; Contra indication to antiemetics; Chronic usage of antiemetics; and Emergent or complicated surgery.

Risk factors for postoperative nausea and vomiting were collected and patients were randomized by cluster into two arms.

Control: No prophylaxis whatever risk score is. Postoperative nausea and vomiting risk factors were not available for practicians.

Intervention: Preoperative collection of postoperative nausea and vomiting risk factors available for practicians. Prophylaxis if risk score is over 2. Prophylaxis of postoperative nausea and vomiting by betamethasone (4mg) and/or droperidol (0.625mg) immediately after cardiac surgery, depending on risk factors in the intervention arm.

All outcomes are assessed at 48 hours of surgery:

Primary: occurrence of postoperative nausea or vomiting Secondary: number of postoperative nausea and vomiting with visual assessment scale (VAS), and antiemetics used for treatment; postoperative pain (VAS) with number of analgesics used; postoperative discomfort (VAS).

Safety data: side effects and QT corrected intervals.

ELIGIBILITY:
Inclusion Criteria:

* Non emergent cardiac surgery
* Age > 18 years
* Affiliation to French Social Security
* Approval of participation to the study

Exclusion Criteria:

* Pregnancy
* Contra indication to antiemetics
* Chronic usage of antiemetics
* Emergent or complicated surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2016-02; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | 48hour
  postoperative nausea and vomiting as a categorical variable

SECONDARY OUTCOMES:
number of postoperative nausea and vomiting | 48hour
postoperative nausea and vomiting (VAS) | 48hour
  Suffering from postoperative nausea and vomiting by visual assessment scale (VAS). VAS is a 100 point scale: 0 indicate absence of nausea or vomiting; 100 indicate maximal nausea and vomiting
postoperative pain (VAS) | 48hour
  VAS is a 100 point scale: 0 indicate absence of pain; 100 indicate maximal pain
postoperative discomfort (VAS) | 48hour
  VAS is a 100 point scale: 0 indicate absence of discomfort; 100 indicate maximal discomfort
Antiemetics (treatment) | 48hour
  Number of antiemetics used as a treatment for postoperative nausea or vomiting
Analgesics | 48hour
  Number of Analgesics used at 48h
Side effects | 48hour
QTc interval | 48hour
  Pre and postoperative QTc (corrected) intervals

CONTACTS AND LOCATIONS:
Locations (1):
- Parly2, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: Yes
On demand